CLINICAL TRIAL: NCT03929705
Title: Assessing the Ability of the T-SPOT®.TB Test to Identify Those at Risk of Active Mycobacterium Tuberculosis Infection Using the Normalized TB Specific Lymphocyte Response
Brief Title: Assessing the Ability of the T-SPOT®.TB Test
Acronym: IQ
Status: Completed | Type: Observational
Sponsor: Oxford Immunotec (Industry)
Responsible Party: Sponsor
Other Study IDs: AF SA 148
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-07

CONDITIONS: Tuberculosis (TB)
Keywords: TB
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PBMCs and plasma will be retained and stored at the Lung Infection and Immunity laboratory Biobank for 3 years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Test Arm 1- T-SPOT.TB assay: T-SPOT.TB test using density gradient isolation (Leucosep) For each subject recruited in the study, cells will be isolated using Leucosep Tubes and T-Cell Xtend reagent according to package insert. For each subject recruited in the study, the T-SPOT.TB assay will be run according to the assay package insert.
- Test Arm 2 -QuantiFERON-TB Gold Plus assay: QuantiFERON-TB Gold Plus, for each subject recruited in the study, the QuantiFERON-TB Gold Plus (QFT-Plus) assay will be run according to the assay package insert.

SUMMARY:
The primary objective of this clinical research study is to demonstrate performance of the normalized TB specific lymphocyte response in identifying patients with active TB disease. The secondary exploratory objective is to demonstrate that active TB cannot be identified using an antigen-to-mitogen ratio derived from an ELISA-based IGRA.

DETAILED DESCRIPTION:
The target number of subjects is 100 active TB and 100 active TB excluded . This study will enroll up to 680 subjects (based on previous enrolment rates of approximately 300-350 subjects enrolled for 50 active TB and 50 active TB excluded).

Study Duration: 6 months

All subjects enrolled in this study will be men or women, aged 18 years or older.

ELIGIBILITY:
Inclusion Criteria: Cohort 1a and 1b

* • Must be at least 18 years of age

  * Must be able to provide informed consent
  * Must be able to provide a minimum of 10 mL of whole blood at each visit (16mL for immunocompromised i.e. HIV+)
  * Must be T-SPOT.TB positive
  * First visit suspect TB subjects with no prior history of TB diagnosis Inclusion Criteria: Cohort 2a and 2b
  * Must be at least 18 years of age
  * Must be able to provide informed consent
  * Must be able to provide a minimum of 10 mL of whole blood at each visit (16mL for immunocompromised i.e. HIV+)
  * Must be T-SPOT.TB positive
  * No prior history of TB diagnosis

Exclusion Criteria: Cohort 1a and 1b

* • Negative in the T-SPOT.TB test

  * Previous or pre-existing confirmed TB diagnosis
  * On anti-TB treatment for more than 1 week*
  * Not meeting inclusion criteria Exclusion Criteria: Cohort 2a and 2b
  * Negative T-SPOT.TB test
  * Previous or pre-existing confirmed TB diagnosis
  * On anti-TB treatment
  * Symptoms of active TB
  * Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and Female 18 years of age and older.
Sampling Method: Non-Probability Sample
Enrollment: 676 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
T-Spot | 6 month study
  The primary objective of this clinical research study is to demonstrate performance of the normalized TB specific lymphocyte response (NTBSLR) in identifying patients with active TB disease. The secondary exploratory objective is to demonstrate that active TB cannot be identified using an antigen-to-mitogen ratio derived from an ELISA-based IGRA.

CONTACTS AND LOCATIONS:
Overall Officials: Keertan Dheda, PhD, Principal Investigator — University of Cape Town
Locations (1):
- University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No